CLINICAL TRIAL: NCT00375206
Title: A Phase I Study to Assess Safety, Tolerability and Immunogenicity of a Trivalent Influenza Vaccine Administered by Particle Mediated Epidermal Delivery (PMED) to Healthy Subjects
Brief Title: A Safety and Immunology Study of a DNA Trivalent Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PM FLS-001
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Influenza
Keywords: PowderMed, DNA vaccine, influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Trivalent DNA Vaccine (PIA0601) with or without DEI-LT (pPJV2012)

SUMMARY:
The purpose of this study is to evaluate how well the vaccine is tolerated at sites where administrations are given and any effects it may have on subjects' wellbeing. The study will also test the ability of vaccine to cause particular immune responses in the body.

DETAILED DESCRIPTION:
Influenza is a contagious disease of the upper airways and the lungs. It rapidly spreads around the world in seasonal epidemics, killing hundreds of thousands of people and having high economic consequences due to healthcare costs and lost productivity. Each year governments recommend groups who are at risk of influenza or its complications to receive influenza vaccination. Current vaccine supply is not sufficient to meet the demand if this recommendation were to be taken up by all. This study is part of the clinical development of a particle mediated epidermal delivery (PMED) trivalent DNA vaccine for the prevention of influenza.This study will investigate the safety and tolerability of this vaccine as well as assess the humoral and cellular immunogenicity of the vaccine in healthy subjects.

ELIGIBILITY:
Ages Eligible for Study:

* 18 Years - 50 Years
* Genders Eligible for Study: Both
* Accepts Healthy Volunteers

Criteria

Inclusion Criteria:

* Healthy adult volunteers (women must be of non child-bearing potential)
* Provided written informed consent

Exclusion Criteria:

* No significant concomitant illness
* No allergy to gold
* No immunosuppression due to disease or treatment
* No previous flu vaccination in 2005 or 2006

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189
Dates: Start 2006-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Safety, tolerability and local reactogenicity - AEs and laboratory parameters

SECONDARY OUTCOMES:
Immunogenicity of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Philip Leese, MD, Principal Investigator — Quintiles, Inc.
Locations (2):
- United States (2):
  - Quintiles Lenexa (QLX), Lenexa, Kansas
  - Biokinetic, Springfield, Missouri